CLINICAL TRIAL: NCT00006398
Title: Randomized, Double-Blind Study of Timolol (A Nonselective Beta-Adrenergic Blocker) vs Placebo to Prevent Complications of Hepatic Portal Hypertension in Patients With Cirrhosis
Brief Title: Prevention of Esophageal Varices by Beta-Adrenergic Blockers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Timolol (completed); R01DK046580 (NIH); YALESM 6618 (Other: Yale School of Medicine); NCT00004641 (obsolete NCT alias)
Record Dates: First submitted 2000-10-05; First posted 2000-10-06 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Esophageal and Gastric Varices; Liver Cirrhosis; Portal Hypertension
Keywords: cirrhosis; esophageal varices; variceal hemorrhage; beta-adrenergic blocker
MeSH Terms: conditions — Esophageal and Gastric Varices; Liver Cirrhosis; Hypertension, Portal; Fibrosis | interventions — Timolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Timolol Maleate (Experimental): Dose titrated from 5 mg per day to up to 80 mg per day depending on heart rate
  Interventions: Drug: Timolol Maleate
- Placebo (Placebo Comparator): Timelol placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Timolol Maleate
  Arms: Timolol Maleate
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to learn whether timolol is useful in preventing or delaying the appearance of gastroesophageal varices, a complication that may develop in the future as a consequence of liver disease. Cirrhosis causes an increased resistance of blood flowing through the liver. This leads to an increased pressure in the portal vein (the vein that takes blood to your liver). High portal pressure is responsible for the appearance of complications of chronic liver disease such as varices and variceal bleeding (bleeding from veins in your esophagus). Timolol belongs to a group of medications called beta-blockers. Beta-blockers decrease high portal pressure and previous studies have shown that beta-blocker pills are useful in preventing bleeding from varices in patients who already have varices. A more desirable effect would be if these pills could prevent not only bleeding from varices but the appearance of varices (and therefore of bleeding).

ELIGIBILITY:
Inclusion Criteria:

* Liver biopsy compatible with cirrhosis.
* Absence of gastroesophageal varices.
* An increased hepatic venous pressure gradient (HVPG) (6mmHg).
* Age over 18 and below 76 years.
* Informed, written consent.
* Absence of exclusion criteria.

Exclusion Criteria:

* Presence of ascites that requires specific treatment (diuretics, paracentesis, peritoneo-venous shunt, etc).
* Proven hepatocellular carcinoma by radiological or histological criteria.
* Splenic or portal vein thrombosis by Doppler-ultrasound.
* Presence of any concurrent disease that is expected to decrease life expectancy to less than one year.
* Patients taking diuretics, beta-blockers, clonidine, prazosin, nitrates, molsidomine and any drug which may have an effect on splanchnic hemodynamics/portal pressure.
* Patients participating in other pharmacological randomized clinical trials.
* Patients with primary biliary cirrhosis and primary sclerosing cholangitis will also be excluded since these entities have a slower progression of the disease, are usually enrolled in other clinical trials and are transplanted at an earlier stage.
* Contraindications to beta-blockers: asthma, COPD with positive broncoconstrictive test, heart failure, A-V block, aortic valve stenosis, organic psychosis, insulin-dependent diabetes, hypersensitivity to beta-blockers.
* Women who are pregnant, nursing or of childbearing potential and who are not using oral or mechanical contraception.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 1993-08 (Actual); Primary Completion 2002-09 (Actual); Study Completion 2002-09 (Actual)

PRIMARY OUTCOMES:
Varices | 6 years
  Development of varices

CONTACTS AND LOCATIONS:
Overall Officials: Roberto J Groszmann, M.D., Principal Investigator — Yale University School of Med.; Norman Grace, M.D. — Tufts University; Jaime Bosch, M.D. — University of Barcelona; Andrew Burroughs, M.D. — University of London; Guadalupe Garcia-Tsao, M.D. — Yale University
Locations (5):
- United States (3):
  - Yale University Sch. of Medicine, New Haven, Connecticut
  - VA CT Healthcare System, West Haven, Connecticut
  - The Faulkner Hospital, Boston, Massachusetts
- Hospital Clinic I Provincial de Barcelona, Barcelona, Catalonia, Spain
- Royal Free Hospital, Hampstead, London, United Kingdom

REFERENCES:
- [Background] Sarin SK, Groszmann RJ, Mosca PG, Rojkind M, Stadecker MJ, Bhatnagar R, Reuben A, Dayal Y. Propranolol ameliorates the development of portal-systemic shunting in a chronic murine schistosomiasis model of portal hypertension. J Clin Invest. 1991 Mar;87(3):1032-6. doi: 10.1172/JCI115062. PMID 1900306
- [Background] Escorsell A, Ferayorni L, Bosch J, Garcia-Pagan JC, Garcia-Tsao G, Grace ND, Rodes J, Groszmann RJ. The portal pressure response to beta-blockade is greater in cirrhotic patients without varices than in those with varices. Gastroenterology. 1997 Jun;112(6):2012-6. doi: 10.1053/gast.1997.v112.pm9178694.
- [Result] Groszmann RJ, Garcia-Tsao G, Bosch J, Grace ND, Burroughs AK, Planas R, Escorsell A, Garcia-Pagan JC, Patch D, Matloff DS, Gao H, Makuch R; Portal Hypertension Collaborative Group. Beta-blockers to prevent gastroesophageal varices in patients with cirrhosis. N Engl J Med. 2005 Nov 24;353(21):2254-61. doi: 10.1056/NEJMoa044456. PMID 16306522
- [Derived] Ripoll C, Groszmann RJ, Garcia-Tsao G, Bosch J, Grace N, Burroughs A, Planas R, Escorsell A, Garcia-Pagan JC, Makuch R, Patch D, Matloff DS; Portal Hypertension Collaborative Group. Hepatic venous pressure gradient predicts development of hepatocellular carcinoma independently of severity of cirrhosis. J Hepatol. 2009 May;50(5):923-8. doi: 10.1016/j.jhep.2009.01.014. Epub 2009 Mar 5. PMID 19303163